CLINICAL TRIAL: NCT05125614
Title: Development of a Staging System and Survival Prediction Model for Advanced Gastric Cancer Patients Without Adjuvant Treatment After Curative Gastrectomy
Brief Title: Gastric Cancer Survival Without Chemotherapy
Status: Completed | Type: Observational
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Ki Bum Park, Clinical Assistant Professor, Saint Vincent's Hospital, Korea
Other Study IDs: apzzap2
Record Dates: First submitted 2021-11-10; First posted 2021-11-18 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Adjuvant chemotherapy; Overall survival; Nomogram; Prediction
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Developement set: Gastric cancer patients who did not receive adjuvant chemotherapy after curative gastrectomy from 2009 to 2016 at Seoul St.Mary's Hospital
  Interventions: Other: No adjuvant chemotherapy
- Validation set: Gastric cancer patients who did not receive adjuvant chemotherapy after curative gastrectomy from 2009 to 2016 at St.Vincent''s Hospital
  Interventions: Other: No adjuvant chemotherapy

INTERVENTIONS:
Other: No adjuvant chemotherapy — There is no intervention differences between 2 groups. We analyzed the data of the patients who did not receive adjuvant chemotherapy.

SUMMARY:
This study is observational study to analyze the actual overall survival of the patients who did not receive adjuvant chemotherapy after curative gastrectomy for gastric cancer.

The investigators developed prediction model for the overall survival of these patients and validated.

DETAILED DESCRIPTION:
Adjuvant chemotherapy (AC) after curative gastrectomy is the standard treatment for patients with locally advanced gastric adenocarcinoma in East Asia; however, for various reasons, some patients do not receive this treatment. The aim of this study was to develop a system that reflects the survival rate of patients without AC. A survival prediction model was developed based on the modified staging system and risk factors for overall survival (OS), which were examined using the Cox proportional hazards regression model. The model was validated for the power of prediction and discrimination, compared with the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th edition; it was externally validated using an independent dataset. the newly developed survival prediction model improves the accuracy of OS prediction for stage II and III gastric cancer patients without AC after curative gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed primary gastric adenocarcinoma
* curative R0 resection with D2 lymph node dissection
* pathologic stage II or III gastric cancer

Exclusion Criteria:

* Patients who received neoadjuvant or AC treatment
* follow-up loss or death within 30 days of surgery
* completion of total gastrectomy
* other malignancy within 5 years before gastrectomy

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Informed consent was not required because of the retrospective nature of the study. For the development set, the database of the Gastric cancer center at Seoul St. Mary's hospital was reviewed between January 2009 and December 2016. The inclusion criteria were: histologically confirmed primary gastric adenocarcinoma, curative R0 resection with D2 lymph node dissection, and pathologic stage II or III. Exclusion criteria were: neoadjuvant or AC treatment, follow-up loss or death within 30 days of surgery, completion of total gastrectomy, and other malignancy within 5 years before gastrectomy. Finally, 185 patients with locally advanced GC, all of whom underwent curative gastrectomy without chemotherapy, were included in the development set. The validation set consisted of patients who satisfied the above inclusion and exclusion criteria from St. Vincent's hospital in the same period. Finally, 157 patients were included in the validation set
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | June-01-2021
  Overall survival of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Ki Bum Park, M.D., Principal Investigator — St Vincent's Hospital
Locations (1):
- Saint Vincent Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol
Time Frame: January 2022, 3 years